CLINICAL TRIAL: NCT04760990
Title: An Open-label Observation Study to Assess the Potential Impact of Disease Modifying Therapies on COVID-19 Outcomes and the Antibody Response Following an Infection With SARS-CoV-2 in Patients With Multiple Sclerosis Within the Swiss Multiple Sclerosis Cohort.
Brief Title: A Study to Assess the Potential Impact of Disease Modifying Therapies on COVID-19 Outcomes and the Antibody Response Following an Infection With SARS-CoV-2 in Patients With Multiple Sclerosis Within the Swiss Multiple Sclerosis Cohort.
Acronym: MS COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Multiple Sclerosis Registry (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02604; me20Mehling
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; COVID-19 (Severe Coronavirus Disease 2019)
Keywords: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); Swiss Multiple Sclerosis Cohort (SMSC)
MeSH Terms: conditions — Multiple Sclerosis; COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — clinical data collection regarding COVID-19 suggestive symptoms or confirmed SARS-CoV-2-infections (medical events), recorded comorbidities (concomitant diseases relevant to MS and COVID-19) and recorded vaccinations (other treatments). This information is systematically collected during the routine clinical visits of the patient within the SMSC every 6-12 months.
Other: analysis of blood samples — analysis of archived serum samples collected every 6-12 months within the SMSC for measurement of anti-SARS-CoV-2 antibodies in pre-pandemic reference samples and prospectively determine the anti-SARS-CoV-2-serostatus during the study period.

SUMMARY:
This nested project of the Swiss Multiple Sclerosis Cohort (SMSC) is to assess the severity of COVID-19 and the magnitude of antibody response after infection with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in patients already treated or not with various immunotherapies for multiple sclerosis followed in the framework of the SMSC.

DETAILED DESCRIPTION:
This nested project of the Swiss Multiple Sclerosis Cohort (SMSC) is to assess the severity of COVID-19 and the magnitude of antibody response after infection with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in patients already treated or not with various immunotherapies for multiple sclerosis followed in the framework of the SMSC.

To assess the frequency and severity of SARS-CoV-2 infections and associated symptoms in the study population, data is collected from systematic questioning during the SMSC-visits and from serum samples collected every 6-12 months within the SMSC (for measurement of anti-SARS-CoV-2 antibodies in pre-pandemic reference samples and prospectively to determine the anti-SARS-CoV-2-serostatus during the study period).

Combining the information on anti-SARS- CoV-2 serostatus and infection history opens the opportunity to determine the number of patients without or with only mild vs. moderate to severe COVID-19 symptoms in large groups of patients with Multiple Sclerosis (MS) treated with immunotherapies targeting various components of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* all patients in the Swiss Multiple Sclerosis Cohort (SMSC)

Exclusion Criteria:

* Patients with Neuromyelitis optica and Radiologically Isolated Syndrome will be excluded
* Existence of a documented refusal of further use of health-related personal data and/or biological material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a nested project within the framework of the SMSC. The SMSC is a prospective multicenter cohort study performed across eight swiss centres. Patients are recruited in the SMSC according to a set of inclusion criteria as specified in the cohort protocol and are only included after a written informed consent is signed.
Sampling Method: Probability Sample
Enrollment: 1181 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of severe COVID-19 as defined by the WHO clinical progression scale (Score 6-9) | through study completion, an average of 3 years
  Incidence of severe COVID-19 as defined by the WHO clinical progression scale (Score 6-9). The WHO clinical progression scale provides a measure of illness severity across a range from 0 (not infected) to 10 (dead). Incidence of severe COVID-19 infections will be assessed by evaluation of collected data on confirmed SARS-CoV-2-infections and their clinical courses.
COVID-19 related death defined by the WHO clinical progression scale (Score 10) | through study completion, an average of 3 years
  COVID-19 related death defined by the WHO clinical progression scale (Score 10) in untreated and treated patients. The WHO clinical progression scale provides a measure of illness severity across a range from 0 (not infected) to 10 (dead).

SECONDARY OUTCOMES:
Proportion of patients with Anti-SARS-CoV-2 seroconversion | through study completion, an average of 3 years
  Proportion of patients with Anti-SARS-CoV-2 seroconversion
Change in mean titers of IgM- and IgG-antibodies against SARS-CoV-2 | through study completion, an average of 3 years
  The Anti-SARS-CoV-2 titer ratios from baseline-samples at pre-pandemic time point to the sample titers during study period will be compared.
Change in individual titers of IgM- and IgG-antibodies against SARS-CoV-2 | through study completion, an average of 3 years
  The Anti-SARS-CoV-2 titer ratios from baseline-samples at pre-pandemic time point to the sample titers during study period will be compared.
Proportion of total confirmed SARS-CoV-2-infections (independent of WHO clinical progression scale Score). | through study completion, an average of 3 years
  Proportion of total confirmed SARS-CoV-2-infections (independent of WHO clinical progression scale Score).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Mehling, PD Dr. med., Principal Investigator — University of Basel, Department of Biomedicine and University Hospital Basel
Locations (7):
- Switzerland (7):
  - Kantonsspital Aarau, Aarau
  - University Hospital Basel, Department of Neurology and Department of Biomedicine, Basel
  - Inselspital Bern, Bern
  - Hôpitaux Universitaires Genève, Geneva
  - Lausanne University Hospital (CHUV), Lausanne
  - Ospedale Regionale di Lugano, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen